CLINICAL TRIAL: NCT06875258
Title: PEnile ReHABilitation After Nerve Sparing Robot-assisted Radical Prostatectomy for Prostate Cancer 2.0, a Multicentre, Randomized Clinical Trial (PEHAB-II)
Brief Title: PEnile ReHABilitation After Nerve Sparing Robot-assisted Radical Prostatectomy for Prostate Cancer 2.0 (PEHAB-II)
Acronym: PEHAB-II
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Antoni van Leeuwenhoek Hospital (Other); Viatris Inc. (Industry); Memidis Pharma (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M23PB2
Record Dates: First submitted 2024-01-08; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Erectile Dysfunction Following Radical Prostatectomy
Keywords: Penile rehabilitation; Vacuum pump device; Sildenafil; Nerve sparing prostatectomy; Quality of life; Sexual quality of life; Prostate cancer survivorship
MeSH Terms: interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intensive rehabilitation arm (Experimental): 12 months daily doses of 75/100 mg Sildenafil combined with vacuum device (VED) therapy for 10 minutes a day, five times a week. Followed by one year on demand use of Phosphodiesterase type 5 inhibitors (PDE5i) (max. 3 times/a week) and/or VED (max. 3 times/a week) and/or Injection therapy (max once/ a week) (based on patients preference and needs).
  Interventions: Drug: Sildenafil; Device: Erectile vacuum device
- Less intensive rehabilitation arm (Active Comparator): Monotherapy with an on-demand dosage of 75/100mg Sildenafil (max. 3 times/a week). Followed by one year on demand use of PDE5i (max. 3 times/a week) and/or VED and/or Injection therapy (max once/ a week). (based on patients preference and needs).
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Sildenafil — Taken daily or on demand. First two weeks dosage of 75mg to manage side effects. If side effects are bearable, dosage will be adjusted to 100mg
  Other Names: Mylan
Device: Erectile vacuum device — 5 days a week, generating 5 erections per day
  Other Names: Active 3 Erection System
  Arms: Intensive rehabilitation arm

SUMMARY:
The PEHAB-II study is prospective, randomized trial designed to assess the effect of two different rehabilitation strategies on the recovery of erectile function in nerve sparing prostatectomy patients. The two rehabilitation strategies consist of 1)12 months daily doses of 100 mg Sildenafil combined with vacuum device (VED) therapy for 10 minutes a day, five times a week or 2) Standard of care: monotherapy with an on-demand dosage of 100mg Sildenafil. The study will be performed in multiple centers in the Netherlands.

DETAILED DESCRIPTION:
Rationale Postoperative erectile dysfunction (ED) is a widely observed side effect of prostate cancer surgery for clinically localized prostate cancer and it has a substantial impact on the quality of life. While nerve-sparing radical prostatectomy (nsRP) has improved the outcomes of erectile function, ED rates remain high even after well-performed nsRP. It is important to note that ED after nsRP is not primarily caused by complete transection (neurotmesis) but rather by neuronal crushing and/or overstretching (neuropraxia) of the neurovascular bundle running alongside the prostate towards the erectile tissue of the penis. It is suggested that the post-operative care is insufficient to consolidate the effects of nsRP because penile rehabilitation is necessary to activate neural recovery as well as to retain the vasculogenic functions of the penile corpora cavernosa. However, the best penile rehabilitation strategy to reduce post-operative ED remains unclear due to a lack of well-designed randomized studies.

Objective This study aims to assess the effect of two different rehabilitation strategies on the recovery rate of ED after nsRP in patients who undergo nsRP.

Main trial endpoint:

The primary endpoint is an adequate, unassisted erection at 24 months after surgery. In this, an adequate unassisted erection is defined as an erection sufficient for successful sexual intercourse without the use of medication or devices. Measured by International Index of Erectile Function - Erectile function domain (IIEF-EF) >/=22 after a one-month drug washout or Expanded Prostate Cancer Index Composite (EPIC) -erection score (sum off Q8b, 9 and 10) >=83 for patients who did not participate in penetrative sex.

Secondary trial endpoints:

Secondary endpoints include erectile function (assisted, unassisted, time to recovery, penile length), health en sexual quality of life (other sexual functions, climacturia, feelings of masculinity, health related quality of life and differences between hetero versus gay/bisexual patients during follow-up), Adherence and side-effects and comparing two sexual function questionnaires.

Trial design This study is a multicentre, randomized, controlled clinical trial.

Trial population:

Patients between the ages of 18- 70 diagnosed with non-metastatic, localized prostate cancer (PCa) who underwent nsRP as primary treatment. A total of 192 patients will be included.

Interventions:

Patients will be randomized 1:1: to arm 1: High intensive therapy using a daily dose of 75-100 mg Sildenafil for 12 month, combined with vacuum device (VED) therapy for 10 minutes a day, five times a week; or to arm 2: Less intensive therapy using 75/100mg Sildenafil on demand (before sexual activity). After these 12 months in therapy, the treatment intensity can be adjusted for the next 12 month until the full neuropraxia recovery time (24 month) has been reached. The treatment option that can be used to intensify the therapy is intracavernosal injection therapy (ICI), in which erections can be obtained quickly by injecting papaverine/phentolamine (Androskat) in the penis. This auxiliary therapy can be an option for those that do not want to wait any longer for the recovery of their spontaneous erections and thus that want to use ICI to obtain erections in the meantime. It is important to note that ICI is not a part of the rehabilitation program and thus is not mandatory. Patients will finish participating in the trial after 24 months follow-up. One month before end of follow-up (23 months) a drug washout will take place.

Endpoints will be assessed after 24 months using validated questionnaires as well and composed validated questions.

Nature and extent of the burden and risks associated with participation, benefit, and group relatedness:

In this study, patients will be evaluated at baseline and every three months thereafter through telephonic appointments, online surveys, and outpatient clinic visits. These outpatient clinic visits will take 20 minutes on average. Patients will fill out HRQoL questionnaires and questionnaires on sexual functioning online. In order to answer these questions correctly, patients will be advised to participate in sexual activity at least once a month. Answering the questionnaires will take approximately 20 minutes. In addition, patients will be asked to provide blood samples once at baseline, to determine testosterone levels, HbA1c, liver enzymes, and lipid profiles. Patients may experience side effects from sildenafil (such as dyspepsia, dizziness, and headache) or the VED (i.e. cold feeling, pain, hematoma, or oedema). These effects are temporary and subside within 25 hours. Participating patients in both arms benefit from free sildenafil and VED, along with the extra attention and guidance provided for sexual recovery, sexual health and erectile function compared to patients that do not participate in the study.

ELIGIBILITY:
Inclusion Criteria:

Pre-screening eligibility criteria

* Age > 18 years and < 70 years
* Patients who have a penis that has developed naturally, without surgical interventions.
* Histologically confirmed PCa
* Scheduled for RP as primary treatment with the intention of at least a one-sided nerve-sparing procedure.
* Non-metastatic disease (cN0M0)
* Pre-operative erections good enough for intercourse (anamnestic)
* Motivated to participate in a penile rehabilitation program

Inclusion criteria

To be eligible to participate in this study, a subject must meet all of the following post- operative criteria:

* All of the above-mentioned pre-screening eligibility criteria
* At least unilateral nerve-sparing or if available Fascia Preservation (FP) score =>5
* A pre-diagnostic anamnestic erection that was good enough for intercourse.
* A pre-diagnostic IIEF-EF>=22 with or without PDE5i. For patients without a partner or did not participate in penetrative sex we use accumulated score of EPIC- erectile function; Q8b, Q9 and Q10 >=83.
* Willing to provide one blood sample to determine testosterone level, hemoglobin 1Ac, liver enzymes and lipid profile
* Testosterone levels of at least >=12 nmol/l, measured pre or post-operative
* A signed informed consent form

Exclusion Criteria:

Pre-screening exclusion criteria:

Regarding history of oncological treatment

* Previous pelvic radiation therapy
* Patients on Androgen Deprivation Therapy (ADT)
* Patients with diseases that affect the red blood cells (e.g., sickle cell anaemia), blood cancer (leukaemia) or bone marrow tumors Regarding history of cardiovascular diseases
* Patients with heart failure New York Heart Association (NYHA) ≥ class 3
* Patients with increased susceptibility to vasodilators include those with left ventricular outflow obstruction (e.g., aortic stenosis, hypertrophic obstructive cardiomyopathy), or those with the rare syndrome of multiple system atrophy manifesting as severely impaired autonomic control of blood pressure.
* Patients with unstable angina pectoris
* Patients using nitride oxide for coronary artery disease
* Patients with hypotension (blood pressure <90/50 mmHg)
* Patients with recent history of stroke or myocardial infarction
* Patients with diseases that affect blood clotting or causes bleeding (i.e. coagulation disorders) or prolonged erections

Other pre-screening exclusion criteria:

* Patients with neurological diseases; such as transient ischemic attack (TIA), Cerebrovascular accident(CVA), Parkinson, and polyneuropathy.
* Allergy regarding Sildenafil
* Patients who have loss of vision in one eye because of non-arteritic anterior ischaemic optic neuropathy (NAION), regardless of whether this episode was in connection or not with previous PDE5 inhibitor exposure.
* Patients with severe hepatic impairment
* Patients with known hereditary degenerative retinal disorders such as retinitis pigmentosa (a minority of these patients have genetic disorders of retinal phosphodiesterases).
* Patients using alpha-blockers, but they may be eligible to participate after discontinuing alpha-blocker use.
* The inability to speak and read in Dutch

Exclusion criteria

* A potential subject who meets any of the following criteria will be excluded from participation in this study:
* All of the above-mentioned pre-screening exclusion criteria
* >pT3b
* Adjuvant radiotherapy or hormonal therapy
* Inability to use VED such as severe penile deformity causing fitting problems

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Erectile function without tools | 24 months
  To determine the difference in rates of patients achieving good unassisted erections at 24 months of follow-up after receiving either 12 months of 75/100mg Sildenafil daily and VED therapy 5 times a week or 75/100mg Sildenafil on demand (≤3 times a week) as a penile rehabilitation program.

SECONDARY OUTCOMES:
Erectile Function | Varying from 6-24 months
  To evaluate time to- and percentage of patients in both arms in regaining unassisted and assisted erectile function sufficient for intercourse during follow-up in each rehabilitation arm. As well to assess and compare stretched penile length at 12 months compared to baseline.
Health en sexual quality of life: | 12 and 24 months
  To compare sexual function scores (i.e. orgasmic function), climacturia, feelings of masculinity, health-related quality of life, partner-interaction, between the treatment groups and between hetero versus gay/bisexual patients during follow-up.
Adherence | 12 months
  To evaluate differences between the groups regarding adherence to the penile rehabilitation program
Best tool to evaluate erectile function: | 6 months
  To evaluate differences in pre-operative IIEF-EF and EPIC-sexual domain scores between patients who are engaged in sexual intercourse and those that are not.
Side effects | 12 months
  To evaluate differences between the groups regarding noted side effects

CONTACTS AND LOCATIONS:
Overall Officials: Inge Cox, MD, Study Director — NCI-Antoni van Leeuwenhoek hospital; Melianthe Nicolai, MD/PhD, Principal Investigator — NCI-Antoni van Leeuwenhoek hospital
Locations (3):
- Netherlands (3):
  - Canisius Wilhelmina Ziekenhuis, Nijmegen, Gelderland
  - Antoni van Leeuwenhoek hospital, Netherlands Cancer Institute, Amsterdam, North Holland
  - Maasstad ziekenhuis, Rotterdam, South Holland

IPD SHARING:
Plan to Share IPD: No